CLINICAL TRIAL: NCT04896034
Title: Evaluation of the Efficacy of the Photobiomodulation on the Pelvi-perineal Pain in Patients in Immediate Post-partum Situation
Brief Title: Efficacy of the Photobiomodulation on the Pelvi-perineal Pain in Immediate Post-partum Situation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PBM study; 2020-A00447-32 (Other: ANSM)
Record Dates: First submitted 2021-04-29; First posted 2021-05-21 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Pelvic Pain
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Intervention Model Description: Single-center, adaptive, prospective, three-arm randomized, controlled, double-blind study for 2 arms.
  3 groups will be constituted, according to a 1:3:3 ratio:
  * 1 group " control 1 " with 2 sessions of PBM ( fake device).
  * 1 experimental group with 2 sessions of PBM (real device)
  * 1 group " control 2 " with standard pain management (i.e. medication).
Who Masked: Participant, Investigator
Masking Description: The experimental group (real device) and the control 1 group ( fake device) will be in double-blind, neither the investigator nor the patient will know the allocated group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- " control 1 " fake MILTA device (Placebo Comparator): Fake device (control 1) which emits 10% red light (and no infrared) so that the difference between the two machines cannot be seen with the naked eye. The magnets present in the real device are absent in the fake machine and replaced by inert materials of the same mass.
  Interventions: Device: " control 1 " fake MILTA device
- MILTA Device (Experimental): The MILTA device used for the study is composed of a panel which gathers 18 emitters composed of red, green and blue LEDs, 3 nanopulsed infrared laser diodes (cold laser), 3 infrared diodes and a permanent magnet
  Interventions: Device: MILTA Device
- " control 2 " standard pain management with medication (No Intervention): In first intention: PARACETAMOL: max 1 g x 4 / 24 h Second intention: IBUPROFEN: max 100 mg x 2 for 48 h Third intention: ACUPAN 20 mg in sugar 3 times per 24 h Last intention: ACTISKENAN 10 mg x 4 / 24 h

INTERVENTIONS:
Device: MILTA Device — Patients in MILTA Device group will each receive 2 sessions of PBM in this study, the first session within 24 hours of delivery, and the second session 24 hours after the first session.
  Arms: MILTA Device
Device: " control 1 " fake MILTA device — Patients in group control 1 will each receive 2 sessions of PBM in this study, the first session within 24 hours of delivery, and the second session 24 hours after the first session.
  Arms: " control 1 " fake MILTA device

SUMMARY:
Photobiomodulation (PBM), evaluated in this study, will be delivered by a CE marked class IIa medical device (MILTA technology), composed of a panel that gathers 18 emitters. This is an innovative, alternative, soft technology, based on a cross action of LED light emission, a low intensity nanopulsed laser and a magnetic tunnel. The sessions last 10 minutes each, in total in the study two sessions will be delivered.

DETAILED DESCRIPTION:
In a woman's life, maternity is an important stage that is not without consequences, not only in daily life but also in future life. Perineal pain syndrome is a problem frequently encountered in the postpartum period and the review of the literature shows that 95 to 100% of women who have given birth by the vaginal way and who present perineal lesions, suffer from perineal pain at 24 hours of the delivery and approximately 60% of them remain painful at 7 days of the delivery. This incidence can decrease to 42% and 11% respectively in the absence of perineal lesions.

Pain in the postpartum period can not only limit a woman's mobility and affect her quality of life, but can also interfere with the care of her child and thus with the establishment of a good mother-child relationship, and thus prevent her from fulfilling her new role as a mother. Finally, acute pain that is not treated can become chronic and affect long-term physical and psychological health.

Pain management in the immediate postpartum period currently involves the use of level 1 analgesics (paracetamol, NSAIDs), the effectiveness of which is uncertain, and level 2 analgesics (weak morphine derivatives, Acupan, Tramadol), which are more effective for pain, but are sometimes badly tolerated or contraindicated in the case of breastfeeding. Recently, several publications tend to show that alternative solutions would allow a more satisfactory approach to the management of painful patients.

In this study, the investigators propose to evaluate the benefit of an innovative analgesic treatment in the immediate postpartum period using photobiomodulation (PBM) by evaluating pain using a Visual Analog Scale. PBM, discovered in the 1950s, uses the properties of light. The PBM corresponds to all the non-thermal and non-cytotoxic biological effects caused by the exposure of tissues to light sources in the visible and near-infrared range. More precisely, certain wavelengths of the light spectrum (red-infrared) lead to a cascade of biological effects within the cell: reduction of pain, regulation of inflammation and acceleration of the healing process.

The objective of this study is to analyze the possibility of replacing chemical medication by a non-invasive, painless technology in patients who have just given birth. This technology is already used for anti-inflammatory and analgesic actions in indications such as stomatology, rheumatology, post-operation and traumatology. This is part of the field of NMIs (non-medicinal interventions).

ELIGIBILITY:
Inclusion Criteria:

* Woman aged 18 years or older
* Primi or multiparous patient
* Natural childbirth, regardless of the method of extraction (spontaneous, vacuum, forceps), and damage to the perineum (simple tear, episiotomy, obstetric anal sphincter injury)
* Patients affiliated to a health insurance plan
* Agreeing to participate in the study and having signed an informed consent

Exclusion Criteria:

* Immediate complications related to the childbirth and requiring management in the continuing care unit (delivery haemorrhage, eclampsia, etc.)
* Severe neonatal complications requiring reanimation.
* Patient with a cardiac pacemaker
* Presence of a disease and/or taking photo-sensitising treatment
* Patient under legal protection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effectiveness of photobiomodulation (PBM) on pain in immediate postpartum patients | 30 minutes after first PBM session for the experimental and control 1 groups
  Evaluated the superiority of the experimental group (MILTA device) to control 1 (fake device) using a Visual Analog Scale (VAS) collected before and after pain management (1st session of PBM)
Evaluation of the effectiveness of photobiomodulation on pain in immediate postpartum patients | 30 minutes after first PBM session for the experimental group or 30 minutes after analgesic treatment for the group control 2
  Evaluated the non-inferiority with of the experimental group (MILTA device) to control 2 (standard of care) using a Visual Analog Scale (VAS) collected before and after pain management

SECONDARY OUTCOMES:
Evaluation of the effectiveness of photobiomodulation on pain after the second PBM session | 30 minutes after second PBM session for the experimental and control 1 groups
  Evaluated the superiority of the experimental group (MILTA device) to control 1 (fake device) using a Visual Analog Scale (VAS) collected before and after pain management (2nd session of PBM)
Characterisation of pain | 30 minutes after first PBM session for the experimental and control 1 groups and 30 minutes after analgesic treatment for the group control 2
  Pain will be characterised using the shortened QDSA questionnaire. The control groups will be compared with the MILTA device.
Characterisation of pain | 30 minutes after second PBM session for the experimental and control 1 groups and 30 minutes after analgesic treatment for the group control 2 (Day 1)
  Pain will be characterised using the shortened QDSA questionnaire. The control groups will be compared with the MILTA device.
Evaluation of the total quantity of analgesics consumed during the hospital stay | through the hospital stay, an average of 2 or 3 days
  Recording of the type and dose of analgesics consumed.
Evaluation of the improvement of postpartum comfort | 30 minutes after first PBM session for the experimental and control 1 groups and 30 minutes after analgesic treatment for the group control 2
  Postpartum confort will be assessed using 5 modalities scale
Evaluation of the improvement of postpartum comfort | 30 minutes after second PBM session for the experimental and control 1 groups and 30 minutes after analgesic treatment for the group control 2 (Day 1)
  Postpartum confort will be assessed using 5 modalities scale
Evaluation of the involvement of caregivers during the hospital stay | through the hospital stay, an average of 2 or 3 days
  Recording the number of calls to the healthcare team related to pain
Safety evaluation | through study completion, an average of 10 days
  Adverse event record

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claude ANTON, MD, Principal Investigator — Clinique la Chataigneraie
Locations (1):
- Clinique la Chataigneraie, Beaumont, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Persico G, Vergani P, Cestaro C, Grandolfo M, Nespoli A. Assessment of postpartum perineal pain after vaginal delivery: prevalence, severity and determinants. A prospective observational study. Minerva Ginecol. 2013 Dec;65(6):669-78. PMID 24346253
- [Background] Morin C, Leymarie MC. La douleur périnéale en post-partum: revue de la littérature. La Revue Sage-femme (2013) 12; 263-268
- [Background] Manresa M, Pereda A, Bataller E, Terre-Rull C, Ismail KM, Webb SS. Incidence of perineal pain and dyspareunia following spontaneous vaginal birth: a systematic review and meta-analysis. Int Urogynecol J. 2019 Jun;30(6):853-868. doi: 10.1007/s00192-019-03894-0. Epub 2019 Feb 15. PMID 30770967
- [Background] Macarthur AJ, Macarthur C. Incidence, severity, and determinants of perineal pain after vaginal delivery: a prospective cohort study. Am J Obstet Gynecol. 2004 Oct;191(4):1199-204. doi: 10.1016/j.ajog.2004.02.064. PMID 15507941
- [Background] Turmo M, Echevarria M, Rubio P, Almeida C. Development of chronic pain after episiotomy. Rev Esp Anestesiol Reanim. 2015 Oct;62(8):436-42. doi: 10.1016/j.redar.2014.10.008. Epub 2014 Dec 30. English, Spanish. PMID 25555717
- [Background] HAS. Douleur chronique: reconnaître le syndrome douloureux chronique, l'évaluer et orienter le patient. Consensus formalisé - December 2008
- [Background] Skovlund E, Fyllingen G, Landre H, Nesheim BI. Comparison of postpartum pain treatments using a sequential trial design. I. Paracetamol versus placebo. Eur J Clin Pharmacol. 1991;40(4):343-7. doi: 10.1007/BF00265841. PMID 2050168
- [Background] Behotas S, Chauvin A, Castiel J, Martin A, Boureau F, Barrat J, Lienhart A. [Analgesic effect of ibuprofen in pain after episiotomy]. Ann Fr Anesth Reanim. 1992;11(1):22-6. doi: 10.1016/s0750-7658(05)80316-8. French. PMID 1443811
- [Background] Gabelle C, Cassa S, Bouvard M, Knoepffler F. Intérêts des anti-inflammatoires non stéroïdes dans les douleurs périnéales du post-partum. J Gyneco. Obst. Biol. Reprod (2004) 33(1): 67 (10)
- [Background] Wehrle M. Prise en charge de la douleur post-épisiotomie en suites de couches: Analyse des pratiques professionnelles à la Maternité Régionale Universitaire de Nancy. Mémoire Université de Lorraine (2015) hal-02110831.
- [Background] Battut A, Nizard J. [Impact of pelvic floor muscle training on prevention of perineal pain and dyspareunia in postpartum]. Prog Urol. 2016 Mar;26(4):237-44. doi: 10.1016/j.purol.2015.09.006. Epub 2015 Oct 9. French. PMID 26455776
- [Background] Golka M. Haute fréquence et douleur périnéale du post-partum. Mémoire Université d'Aix Marseille (2017) dumas-01646228
- [Background] Boureau F, Luu M. Méthodes d'évaluation de la douleur. Douleur et Analgésie (1988) 6; 1(2): 65-78.
- [Background] Hamblin MR. Mechanisms and applications of the anti-inflammatory effects of photobiomodulation. AIMS Biophys. 2017;4(3):337-361. doi: 10.3934/biophy.2017.3.337. Epub 2017 May 19. PMID 28748217
- [Background] Moreira Rocha Jr A. Et al. Effects of Low-Level Laser Therapy on the progress of wound healing in humans: the contribution of in vitro and in vivo experimental studies. J. Vas. Bras 2007; 6(3): 258-266
- [Background] Luo L, Sun Z, Zhang L, Li X, Dong Y, Liu TC. Effects of low-level laser therapy on ROS homeostasis and expression of IGF-1 and TGF-beta1 in skeletal muscle during the repair process. Lasers Med Sci. 2013 May;28(3):725-34. doi: 10.1007/s10103-012-1133-0. Epub 2012 Jun 20. PMID 22714676
- [Background] Cidral-Filho FJ, Mazzardo-Martins L, Martins DF, Santos AR. Light-emitting diode therapy induces analgesia in a mouse model of postoperative pain through activation of peripheral opioid receptors and the L-arginine/nitric oxide pathway. Lasers Med Sci. 2014 Mar;29(2):695-702. doi: 10.1007/s10103-013-1385-3. Epub 2013 Jul 6. PMID 23832179
- [Background] Enwemeka CS, Parker JC, Dowdy DS, Harkness EE, Sanford LE, Woodruff LD. The efficacy of low-power lasers in tissue repair and pain control: a meta-analysis study. Photomed Laser Surg. 2004 Aug;22(4):323-9. doi: 10.1089/pho.2004.22.323. PMID 15345176
- [Background] Ahangar FA et Al. Efficace of nano-pulsed magneto infrared Laser Therapy with a fixed dose combination tablet of oral Ibuprofen and paracetamol on the reduction of endodontie pain: a clinical study. Contemporary Med. Res. (2017); 4(8): 1782-1787
- [Background] Chow RT, Johnson MI, Lopes-Martins RA, Bjordal JM. Efficacy of low-level laser therapy in the management of neck pain: a systematic review and meta-analysis of randomised placebo or active-treatment controlled trials. Lancet. 2009 Dec 5;374(9705):1897-908. doi: 10.1016/S0140-6736(09)61522-1. Epub 2009 Nov 13. PMID 19913903
- [Background] Ezzati K, Fekrazad R, Raoufi Z. The Effects of Photobiomodulation Therapy on Post-Surgical Pain. J Lasers Med Sci. 2019 Spring;10(2):79-85. doi: 10.15171/jlms.2019.13. Epub 2019 Feb 25. PMID 31360374
- [Background] FDA, Multiple Endpoints in Clinical Trials Guidance for Industry, January 2017